CLINICAL TRIAL: NCT04389931
Title: Effect of Omega 3 as an Immunomodulator Adjunct to Periodontal Debridement: A Randomized Controlled Clinical Trial
Brief Title: Effect of Omega 3 as an Immunomodulator Adjunct to Periodontal Debridement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Responsible Party: Principal Investigator, Mariely Navarrete, Associate Professor, Faculty of Dentistry Andres Bello University, Viña del Mar campus, Universidad Nacional Andres Bello
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 047
Record Dates: First submitted 2020-05-10; First posted 2020-05-15 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Periodontitis
Keywords: Fatty Acids, Omega-3; Periodontal debridement; Immunomodulation; Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Lactose; Docosahexaenoic Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized controlled trial, where patients with a history of Moderate Periodontitis with moderate rate of progression (Stage II grade B) and Severe Periodontitis with potential for additional tooth loss and moderate rate of progression (Stage III grade B). The intervention group received nonsurgical periodontal therapy (SRP) plus Omega 3, and the control group received SRP plus placebo. The clinical variables were measured before the treatment, the first, third and six month of the end of the SRP, while the microbiological variables were measured before the treatment and in the third month after treatment.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontal treatment, lactose tab (Placebo Comparator): Periodontal treatment (scaling and root planning) and two tablets containing lactose once a day for 90 days immediately after the scaling and root planning.
  Interventions: Other: Lactose tab
- Periodontal treatment, Omega 3 (Experimental): Periodontal treatment (scaling and root planning) and two tablets containing 1g of Omega 3 once a day for 90 days immediately after the scaling and root planning.
  Interventions: Drug: Omega 3

INTERVENTIONS:
Other: Lactose tab — Two tablets containing lactose Procedure: Periodontal treatment Scaling and root planning
  Arms: Periodontal treatment, lactose tab
Drug: Omega 3 — Two tablets containing 1g Omega 3. Procedure:Periodontal treatment Scaling and root planning
  Other Names: Omega 3 fatty acid
  Arms: Periodontal treatment, Omega 3

SUMMARY:
This study evaluates the effect of the systemic administration of Omega 3 as a therapy associated with non-surgical periodontal treatment, in the clinical and microbiological variables of patients with Moderate Periodontitis with moderate rate of progression (Stage II grade B) and Severe Periodontitis with potential for additional tooth loss and moderate rate of progression (Stage III grade B). A double-blind, randomized, controlled trial was conducted with 18 voluntary patients with a history of moderate to severe chronic periodontitis, who met the inclusion and exclusion criteria and signed an informed consent. The intervention group received Scaling and Root Planning (SRP) plus Omega 3, and the control group received SRP plus placebo. Probing depth (PD), Clinical Attachment Level (CAL), Biofilm Index (BI) and Bleeding on Probing (BOP) were evaluated as clinical variables while Porphyromonas gingivalis (Pg), Tannerella forsythia (Tf), Treponema denticola (Td), Fusobacterium nucleatum (Fn) were the microbiological variables detected by conventional Polymerase chain reaction (PCR).

DETAILED DESCRIPTION:
Definition of the sample: Patients over 18 years old admitted to the Diagnostic Unit of the Faculty of Dentistry (DUFD), Viña del Mar campus of the University National Andres Bello (UNAB) during 2016, with a diagnosis of moderate or severe chronic periodontitis, meeting both the inclusion and exclusion criteria and voluntarily agree to participate of the present research work, signing an informed consent. The chosen participants were informed of the nature of the research, potential risks and compensation for participating in the study, obtaining informed consent from every patient. Sample Size Calculation: To calculate the minimum sample size necessary for the constitution of the control and intervention groups, the variance of the probing depth difference were considered as fixed values, which were based on the results described above.Considering the above and using a level of significance of 5%, a statistical power of 80% and an estimation error of 1 mm, at least 7 patients were obtained for each group, giving a total of 14 minimum subjects to study. Protocol and clinical exam: Out of a total of 31 patients who were selected, 20 of those who met the inclusion criteria were randomly assigned by the study coordinator to one of the two groups using a random generation sequence employing a software. Two subjects declined to participate in the research. In this way, two groups were formed to investigate: an intervention group (8 subjects) that received SRP plus 2 g of a Omega once a day for 90 days immediately after the SRP, and a control group (10 subjects) that received SRP plus placebo under the same conditions as the intervention group. One subject of the control group and two of intervention, were lost during the six month control. Finally, fifteen patients entering the study also completed it. No compliance problems were noted, all patients followed the protocol of the study. None subjects reported specific adverse effects.

Randomization: Only the main investigator, who made the randomization by using the Epidat 4.0 program, had knowledge about the content of the containers and the group to which each patient belonged in the study, therefore, was in charge of labeling the containers, achieving in this way that collaborators and participants in the investigation did not know their content until after the study was finished. Standardization and calibration: The data was collected using instruments and supplies with the same commercial brands, in a single chair, under the same lighting and by a single examiner in the case of clinical data and another examiner for microbiological variables. The complete process of PCR was performed by a biochemist belonging to the microbiology laboratory, Santiago campus of the UNAB. An interexaminer calibration was performed, where the only clinical examiner was calibrated by a specialist in periodontics, recording the data obtained in a calibration sheet. For this, a minimum of 10 subjects were evaluated, in which a site of one tooth belonging to each quadrant was randomly selected. Periodontopathogens: The presence of periodontopathogens was considered when exposing the agarose gel of the electrophoresis to ultraviolet light, a band at the site of the 197 base pairs (bp) was observed in the lane possessing the patient's subgingival bioflora sample of Pg, 316 base pairs for Td, 745 for Tf and 167 for Fn. Data collection and instrument: Prior to the data collection, all subjects belonging to the study were asked for a panoramic radiograph for diagnostic purposes. Subsequently, the periodontal examination was performed registering the clinical variables described above in a clinical record. Obtaining microbiological samples: The microbiological examination was performed before SRP on both groups. The collection of microbiological samples was based on a protocol that is used at the University of Chile. Using sterile paper cones number 40, a sample of subgingival biofilm was taken from the site with the highest CAL, within those with PD ≥ 5mm, and an oral hygiene instruction was performed. Before the collection of subgingival biofilm, the area was cleaned with a sterile gauze to eliminate the supragingival biofilm. Then, with a tweezer, a paper cone was taken, and its tip was placed in the sulcus of the study site for 20 seconds, to ensure the absorption of the crevicular fluid and subgingival biofilm. Each biological sample obtained was suspended in an Eppendorf tube with 1 ml of distilled water and transported in a refrigerator at a temperature of 4°C approximately, within a time not exceeding 3 hours, to be then temporarily stored at -80°C, until its transfer and subsequent extraction of deoxyribonucleic acid (DNA) and PCR technique processing. The time between sampling and DNA extraction did not exceed 48 hours, to avoid deterioration of the biological material. Periodontal Treatment: Once the preliminary collection of all the variables was completed, non-surgical periodontal treatment was carried out, beginning with supra and subgingival full-mouth decontamination, using an electric piezo (DTE®, Guilin Woodpecker Medical Instrument Co., Ltd., Guilin, Guangxi , People's Republic of China), followed by root planning at sites presenting PD ≥ 5mm and CAL≥ 4mm, using Gracey curettes (Hu-Friedy® Manufacturing Inc., Chicago, Illinois (IL), USA). This therapy was performed in all patients, both in the intervention and control group, under full mouth treatment protocol, in 1 or 2 work sessions, lasting from 1 to 2 hours, achieving treatment within 24 hours. Omega 3 or placebo administration: At the end of the last treatment session, the Omega 3 (Omega 3, Galenic Pharmacy) or a placebo (Lactose, Galenic Pharmacy) was administered, depending on the group, intervention or control respectively, to which the patient belonged. For both therapies, the administration regimen was 2 tablets of 1g orally per day, for 90 consecutive days.To maintain the double-blind, the containers used for the Omega 3 and placebo presented the same characteristics regarding size and color. About the Omega 3 tablets and placebo, these were visually identical. Subsequently, at the first, third and six month after the end of the nonsurgical treatment, a new collection of all the clinical variables measured at the beginning of the study was performed, while the microbiological variables were measured again at the third month after treatment, from the same site used in the first sampling.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years.
* Patients American Society of Anesthesiologists (ASA) I or ASA II compatible with local anesthesia procedures.
* Present at least 10 natural teeth, excluding semi-erupted third molars.
* Present at least 6 sites with a probing depth (PD) ≥ 5mm and clinical attachment loss (CAL) ≥ 4mm

Exclusion Criteria:

* Patients with hemostasis disorders.
* Patients who use any medication associated with gingival disorders such as: Anticonvulsants (Phenytoin), Calcium channel blockers (Nifedipine), Immunosuppressive drugs (Cyclosporins).
* Patients with systemic diseases that affect the immunoinflammatory response.
* Patients under treatment with antacids on a regular basis due to chronic gastritis and / or self-medication with antacids.
* Patients under treatment with drugs such as: warfarin, digoxin and acetylsalicylic acid.
* Previous history of allergy to local anesthetics.
* Patients presenting orthodontic appliances.
* Patients who have received antibiotic treatment in the last 3 months.
* Patients who have received periodontal treatment.
* Pregnancy.
* Carriers of valvular prostheses or failures in heart valves, with endocarditis risk.
* Patients who are physically and intellectually incapacitated to participate, according to chilean law number 20,584, title II, paragraph 8, article 28.
* Heavy smoking patients, which is smoking more than 10 cigarettes per day.
* Patients allergic to Omega 3 or seafood or its derivatives: fish, shellfish, algae, etc.
* Patients with lactose intolerance.

Ages: 39 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Difference between groups for the mean of sites with Probing depth (PD) ≤ 3 mm, PD ≥ 4 mm and PD ≥ 7 mm in stage II or III grade B periodontitis patients, before and 1, 3 and 6 month after SRP with placebo or Omega 3. | Baseline,1,3 and 6 month.
  Before, 1, 3 and 6 month after performing SRP with placebo or Omega 3, PD was measured in all the patients in the study and corresponds to the distance in millimeters from the gingival margin (MG) to the inserted probe´s tip of the most apical portion of the periodontal pocket. It was obtained by measuring with a North Carolina periodontal probe (Hu-Friedy® Manufacturing Inc., Chicago, IL, USA), from the bottom of the pocket to the MG, in a position parallel to the vertical axis of the tooth, with a pressure no greater than 0.25 Newton (N). PD was performed in a circular direction over the entire surface of each tooth, registering the 6 deepest sites per tooth (mesiobuccal, buccal, distobuccal,distolingual, lingual and mesiolingual). Subsequently, those sites with PD ≥ 3 mm, PD ≥ 4 mm, PD ≥ 7 mm were counted and the student t test was applied to observe if there were significant differences between both treatment groups.

SECONDARY OUTCOMES:
Risk for disease progression, according to Lang & Tonetti (2003). | Baseline and 6 month.
  Percentage of subjects presenting low (≤ 4 sites with PD ≥ 5 mm),moderate (5-8 sites with PD ≥ 5 mm) or high (≥ 9 sites with PD ≥5 mm), before and 6 month after performing SRP with placebo or Omega 3.
Clinical Attachment Level (CAL) gain in the sixth month after SRP with placebo or Omega 3. | Baseline and 6 month.
  Before and 6 month after performing SRP, CAL was measured in all the patients in the study and corresponds to the distance measured in millimeters from the cementum enamel junction to the tip of the probe inserted to the most apical portion of the periodontal pocket. It was obtained using a North Carolina periodontal probe (Hu-Friedy® Manufacturing Inc., Chicago, IL, USA), in a position parallel to the vertical axis of the tooth, with a pressure not greater than 0.25 N.
Difference between groups for the Biofilm Index (BI) ,in stage II or III grade B periodontitis patients before and 1, 3 and 6 month after performing SRP with placebo or Omega 3. | Baseline,1, 3 and 6 month.
  Before,1,3 and 6 month after performing SRP, BI was measured in all the patients in the study. BI is percentage of dental surfaces with staining, through the use of biofilm developers. To obtain the index, a curaprox developer tablet was dissolved in a plastic cup with water and with a cotton ball this solution was applied on all of the tooth surfaces, recording only those that were stained. The calculation was made by dividing the surfaces that stained by the total surfaces, which corresponds to the number of teeth present multiplied by 4, and multiplying this value by 100. Subsequently, student t test was applied to observe if there were significant differences between both treatment groups.
Difference between groups for the bleeding on probing (BOP) Index, in stage II or III grade B periodontitis patients before and 1, 3 and 6 month after performing SRP with placebo or Omega 3. | Baseline,1, 3 and 6 month.
  Before,1, 3 and 6 month after performing SRP, BOP was measured in all the patients in the study. BOP is the percentage of sites that bleed when probing. It was recorded during PD measurement with a North Carolina periodontal probe (Hu-Friedy® Manufacturing Inc., Chicago, IL, USA) and was considered positive if it occurs 20 seconds after probing. The calculation was made by dividing the sites that bled by the total sites, which corresponds to the number of teeth present multiplied by 6, and multiplying this value by 100. Subsequently, student t test was applied to observe if there were significant differences between both treatment groups.
Presence of periodontopathogens before, 3 and 6 month after performing SRP with placebo or Omega 3. | Baseline, 3 and 6 month.
  Before, 3 and 6 month after performing SRP, the microbiological examination was performed on both groups. The biofilm samples were analyzed to detect the presence of four bacterial species: Porphyromonas gingivalis (Pg),Tannerella forsythia (Tf), Treponema denticola (Td), Fusobacterium nucleatum (Fn) by Polymerase chain reaction(PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Mariely A Navarrete, MSc, Study Director — Universidad Nacional Andres Bello; Mariely A Navarrete Riffo, MSc, Principal Investigator — Universidad Nacional Andres Bello
Locations (1):
- Universidad Nacional Andres Bello, Viña del Mar, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Background] Meissner K, Bingel U, Colloca L, Wager TD, Watson A, Flaten MA. The placebo effect: advances from different methodological approaches. J Neurosci. 2011 Nov 9;31(45):16117-24. doi: 10.1523/JNEUROSCI.4099-11.2011. PMID 22072664
- [Background] Suchy FJ, Brannon PM, Carpenter TO, Fernandez JR, Gilsanz V, Gould JB, Hall K, Hui SL, Lupton J, Mennella J, Miller NJ, Osganian SK, Sellmeyer DE, Wolf MA. National Institutes of Health Consensus Development Conference: lactose intolerance and health. Ann Intern Med. 2010 Jun 15;152(12):792-6. doi: 10.7326/0003-4819-152-12-201006150-00248. Epub 2010 Apr 19. No abstract available. PMID 20404261
- [Background] Jellema P, Schellevis FG, van der Windt DA, Kneepkens CM, van der Horst HE. Lactose malabsorption and intolerance: a systematic review on the diagnostic value of gastrointestinal symptoms and self-reported milk intolerance. QJM. 2010 Aug;103(8):555-72. doi: 10.1093/qjmed/hcq082. Epub 2010 Jun 3. PMID 20522486
- [Result] Lang NP, Tonetti MS. Periodontal risk assessment (PRA) for patients in supportive periodontal therapy (SPT). Oral Health Prev Dent. 2003;1(1):7-16. PMID 15643744
- [Result] Van Dyke TE, Hasturk H, Kantarci A, Freire MO, Nguyen D, Dalli J, Serhan CN. Proresolving nanomedicines activate bone regeneration in periodontitis. J Dent Res. 2015 Jan;94(1):148-56. doi: 10.1177/0022034514557331. Epub 2014 Nov 11. PMID 25389003
- [Result] Deore GD, Gurav AN, Patil R, Shete AR, Naiktari RS, Inamdar SP. Omega 3 fatty acids as a host modulator in chronic periodontitis patients: a randomised, double-blind, palcebo-controlled, clinical trial. J Periodontal Implant Sci. 2014 Feb;44(1):25-32. doi: 10.5051/jpis.2014.44.1.25. Epub 2014 Feb 26. PMID 24616831